CLINICAL TRIAL: NCT06797765
Title: Optical Coherence Tomography Angiography in Neurological Disease: A Pilot Study
Brief Title: Optical Coherence Tomography Angiography in Neurological Disease
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Noah Jouett, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-0876
Record Dates: First submitted 2024-12-21; First posted 2025-01-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Octa; Stroke; Subarachnoid Hemorrhage; Intracerebral Hemorrhage
MeSH Terms: conditions — Stroke; Subarachnoid Hemorrhage; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Normal healthy human subjects
  Interventions: Device: OCTA
- Patients: Patients with neurological disease
  Interventions: Device: OCTA

INTERVENTIONS:
Device: OCTA — Optical Coherence Tomography Angiography

SUMMARY:
Optical Coherence Tomography Angiography (OCTA) is a non-invasive tool that images the neurovascular structures of the eye by using near-infrared light. Previous literature has demonstrated the potential of OCTA as a screening tool in stroke, but its utility in other neurological illness such as intracranial hemorrhage is unclear. Hence, this pilot study will gather preliminary data to support future grant applications to investigate this area more fully by recruiting patients with neurological illness and healthy controls and comparing their OCTA imaging parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient admitted to the neuroscience intensive care unit with a diagnosis of: subarachnoid hemorrhage, intracerebral hemorrhage, intracranial aneurysm (ruptured or unruptured), intracranial vascular malformation, ischemic stroke, seizure disorder, intracranial infection, intracranial tumor(s), inflammatory demyelinating disease, traumatic brain injury and/or neuromuscular respiratory failure OR subjects from the community without major neurologic, cardiovascular, pulmonary or metabolic disease

Exclusion Criteria:

* Pregnancy
* Non-English speaking
* GCS motor score less than 6 (i.e. must be able to follow commands)
* Temporary or permanent physical limitation that renders the patient unable to sit up and look inside OCTA device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Control and Patient population
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Vascular and Perfusion Density in healthy controls | Once (approx. 10 mins)
  Quantitative measure of retinal microperfusion. No definite time points are defined since different neurological diseases have different patterns of evolution and patient/provider availability may change.
Vascular and Perfusion Density in Patients with neurological disease | Throughout study completion up to 28 days
  Quantitative measure of retinal microperfusion. No definite time points are defined since different neurological diseases have different patterns of evolution and patient/provider availability may change.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Pilot study

REFERENCES:
- [Background] Patton N, Aslam T, Macgillivray T, Pattie A, Deary IJ, Dhillon B. Retinal vascular image analysis as a potential screening tool for cerebrovascular disease: a rationale based on homology between cerebral and retinal microvasculatures. J Anat. 2005 Apr;206(4):319-48. doi: 10.1111/j.1469-7580.2005.00395.x. PMID 15817102